CLINICAL TRIAL: NCT02039427
Title: The Effect of Prophylactic Ketorolac on Sore Throat After Thyroid Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeungnam University College of Medicine (Other)
Responsible Party: Principal Investigator, Sung Mee Jung, M.D., Yeungnam University College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: YUH-3368-sore throat
Record Dates: First submitted 2014-01-15; First posted 2014-01-17 (Estimated); Results first posted 2017-07-31 (Actual); Last update posted 2017-08-28 (Actual); Status verified 2017-07

CONDITIONS: Anesthesia Intubation Complication; Tracheal Disease
Keywords: Sore throat; Hoarseness; Intubation; Thyroidectomy; Ketorolac; Dexamethasone
MeSH Terms: conditions — Tracheal Diseases; Pharyngitis; Hoarseness | interventions — Ketorolac; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Normal saline(Placebo) 2 ml 5 min before induction Normal saline 2 ml 10 min before end of surgery
  Interventions: Drug: Placebo
- Preketorolac (Active Comparator): Ketorolac 30 mg 5 min before induction Normal saline 2 ml 10 min before end of surgery
  Interventions: Drug: Ketorolac
- Postketorolac (Active Comparator): Normal saline 2 ml 5 min before induction Ketorolac 30 mg 10 min before end of surgery
  Interventions: Drug: Ketorolac
- Dexamethasone (Active Comparator): Dexamethasone 10 mg (total volume 2 ml) 5 min before induction Normal saline 2 ml 10 min before end of surgery
  Interventions: Other: Dexamethasone

INTERVENTIONS:
Drug: Ketorolac — ketorolac 30 mg mixed with normal saline 1 ml : total volume of 2 ml
  Other Names: Kerola
  Arms: Postketorolac; Preketorolac
Other: Dexamethasone — dexamethasone acetate10 mg : total volume of 2 ml
  Arms: Dexamethasone
Drug: Placebo — Normal saline 2 ml
  Other Names: control
  Arms: Placebo

SUMMARY:
Sore throat is one of most frequent complaints related to general anesthesia with tracheal intubation. Although sore throat is regarded as a minor and short-lasting discomfort after surgery, its incidence and intensity in high risk patients such as female gender, head and neck surgery and difficult laryngoscopy or intubation may attribute to prolong postoperative recovery and give patient dissatisfaction.

Even though the pathophysiology of post-intubation airway symptoms is not completely clarified yet, the mucosal damage related inflammation at the cuff of endotracheal tube has been thought to be an essential trigger. Thus anti-inflammatory medication has been commonly used strategy to prevent postoperative airway discomfort after intubation. The preoperative administration of dexamethasone has been reported to reduce the incidence and severity of postoperative sore throat, but it is accompanied with the adverse effects such as hyperglycemia, delayed wound healing and increased infection in surgical patients. Ketorolac, non-steroidal anti-inflammatory drug (NSAID), is an analgesic that commonly used for postoperative pain control and has anti-inflammatory effect.

Therefore, the investigator designed to evaluate the effect of ketorolac on sore throat in comparison to dexamethasone after thyroidectomy in female adult patients

DETAILED DESCRIPTION:
Ketorolac, NSAID, has not been evaluated as a pharmacologic strategy to reduce postoperative sore throat yet. The investigator will explore how the analgesic and anti-inflammatory effects of ketorolac influence airway symptoms following general anesthesia with tracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

1. American society of Anesthesiologists(ASA) physical status 1 and 2
2. 20-60 years old female
3. elective scheduled thyroidectomy

Exclusion Criteria:

surgery longer than 3 hours Previous history of or expected difficult tracheal intubation Laryngoscope grade (by Cormack and Lehane) of 3 or 4 2 more trial for intubation BMI > 30 Hypersensitivity to ketorolac history of asthma respiratory tract infection during the past 6 weeks Renal dysfunction (creatinine > 1.5 mg/dl or oligouria) Hepatic dysfunction (ALT :> 50% more than normal value) Use of corticosteroid, NSAIDS, angiotensin converting enzyme in 10 days Medication for gastritis, gastric ulcer Upper gastrointestinal bleeding history Diabetes mellitus

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 192 (Actual)
Dates: Start 2014-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sung Mee Jung, M.D., Principal Investigator — Yeungnam University College of Medicine
Locations (1):
- Yeungnam University Hospital, Daegu, South Korea

REFERENCES:
- See also: Complaints of sore throat after tracheal intubation: a prospective evaluation — http://www.ncbi.nlm.nih.gov/pubmed/15892411
- See also: Gender differences in risk factors for airway symptoms following tracheal intubation — http://www.ncbi.nlm.nih.gov/pubmed?linkname=pubmed_pubmed&from_uid=15892411
- See also: Dexamethasone for preventing postoperative sore throat: a meta-analysis of randomized controlled trials — http://www.ncbi.nlm.nih.gov/pubmed/24357270

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted Yeungnam University Hospital in South korea from Oct. 2013 to Oct. 2015. One hundred and ninety - two female adults aged between 20 and 65 years, ASA physical status I or II scheduled for elective primary thyroidectomy under general anesthesia were enrolled.
Pre-assignment Details: Patients with a airway problem, recent upper respiratory tract infection, obese, inflammation or hemorrhage in the upper gastrointestinal tract, use of NSAID or steroid medication, allergy to the general anesthetic used in this study were excluded.
Groups:
- Placebo: Normal saline(Placebo) 2 ml at 5 min before induction and Normal saline(Placebo) 2 ml at 10 min before end of surgery
  Placebo: Normal saline 2 ml
- Preketorolac: Ketorolac 30 mg at 5 min before induction and Normal saline(Placebo) 2 ml at 10 min before end of surgery
  Ketorolac: ketorolac 30 mg mixed with normal saline 1 ml : total volume of 2 ml
- Postketorolac: Normal saline(Placebo) 2 ml at 5 min before induction and Ketorolac 30 mg at 10 min before end of surgery
  Ketorolac: ketorolac 30 mg mixed with normal saline 1 ml : total volume of 2 ml
- Dexamethasone: Dexamethasone 10 mg at 5 min before induction and Normal saline(Placebo) 2 ml at 10 min before end of surgery
  Dexamethasone: dexamethasone acetate 10 mg mixed with normal saline : total volume of 2 ml
Period: Overall Study
Arm/Group | Placebo | Preketorolac | Postketorolac | Dexamethasone
Started | 48 | 48 | 48 | 48
Completed | 45 | 47 | 45 | 43
Not Completed | 3 | 1 | 3 | 5
Not completed — Duration of surgery > 3h | 1 | 1 | 0 | 0
Not completed — Withdrawal on concent | 0 | 0 | 0 | 1
Not completed — Cancellation of surgery | 0 | 0 | 1 | 0
Not completed — Loss of follow - up | 1 | 0 | 2 | 4
Not completed — Steroid Use | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Preketorolac | Postketorolac | Dexamethasone | Total
Number analyzed (Participants) | 45 | 47 | 45 | 43 | 180
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 45 | 47 | 45 | 43 | 180
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.2 (10.1) | 49.5 (9.2) | 47.3 (9.3) | 46.0 (11.1) | 47.8 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 47 | 45 | 43 | 180
  Male | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of Postoperative Sore Throat(POST) Using Ketorolac and Dexamethasone in Womend After Thyroidectomy
Description: The investigator asked scales to patients at 1, 6 and 24h after extubation. POST was defined as discomfort at larynx or pharynx at rest and during swallowing after surgery and was assessed using a 4-grade scale (0-3) based on verbal responses to questions: 0, none; 1, mild (less severe than with a cold); 2, moderate (similar with a cold); 3 severe (more severe than with a cold)
  ● Incidence of sore throat : if patient rates sore throat scale more than 1, investigator will record as positive symptom.
Time Frame: at 1, 6 and 24 hours after thyroidectomy
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Preketorolac | Postketorolac | Dexamethasone
Number analyzed (Participants) | 45 | 47 | 45 | 43
Participants
  Sore throat Rest at 1h | 43 | 44 | 42 | 41
  Sore throat Rest at 6h | 32 | 34 | 33 | 25
  Sore throat Rest at 24h | 20 | 21 | 25 | 15
  Sore throat Swallowing at 1h | 44 | 45 | 44 | 42
  Sore throat Swallowing at 6h | 44 | 42 | 40 | 35
  Sore throat Swallowing at 24h | 42 | 37 | 37 | 29

2. Secondary Outcome: The Incidence of Postoperative Hoarseness(PH) Using Ketorolac and Dexamethasone in Womend After Thyroidectomy
Description: The investigator asked scales to patients at 1, 6 and 24h after extubation. PH was assessed using a 4-grade scale (0-3): 0, none; 1, mild (noticed by the patient only); 2, severe (obvious to observer); 3 aphonia (silence of voice)
  ● Incidence of hoarseness: If patient exhibit hoarseness scale more than 1, investigator will record as positive sign
Time Frame: at 1, 6 and 24 hours after thyroidectomy
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Preketorolac | Postketorolac | Dexamethasone
Number analyzed (Participants) | 45 | 47 | 45 | 43
Participants
  Hoarseness at 1h | 42 | 44 | 40 | 40
  Hoarseness at 6h | 37 | 36 | 39 | 35
  Hoarseness at 24h | 34 | 28 | 29 | 22

3. Other Pre Specified Outcome: Potential Side Effects Associated With the Study Drugs
Description: Potential side effects associated with the study drugs, such as anlgesic use, nausea and vomiting.
Time Frame: at 1, 6 and 24 hours after extubation
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Preketorolac | Postketorolac | Dexamethasone
Number analyzed (Participants) | 45 | 47 | 45 | 43
Participants
  Analgesic use at 1h | 14 | 4 | 6 | 9
  Analgesic use at 6h | 2 | 0 | 0 | 0
  Analgesic use at 24h | 1 | 0 | 0 | 0
  Nausea at 1h | 10 | 11 | 13 | 15
  Nausea at 6h | 2 | 7 | 6 | 1
  Nausea at 24h | 0 | 1 | 2 | 0
  Vomiting at 1h | 0 | 2 | 1 | 1
  Vomiting at 6h | 0 | 2 | 1 | 0
  Vomiting at 24h | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1h, 6h and 24h after surgery
Arm/Group | Placebo | Preketorolac | Postketorolac | Dexamethasone
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/47 | 0/45 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/47 | 0/45 | 0/43
Other Adverse Events (participants affected / at risk) | 0/45 | 0/47 | 0/45 | 0/43

LIMITATIONS AND CAVEATS:
The present study has some limitations. First, the dose of dexamethasone and ketorolac may not be equipotent in terms of anti-inflammatory efficacy. Second, postoperative pain control might affect the incidence and severity of the POST.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No